CLINICAL TRIAL: NCT03524313
Title: Assessment of Cardiac Output With End-tidal Carbon Monoxide
Brief Title: Assessment of Cardiac Output With EtCO2
Acronym: COCO2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2018/367
Record Dates: First submitted 2018-04-09; First posted 2018-05-14 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2019-12

CONDITIONS: Cardiac Output
Keywords: cardiac output; end tidal carbon monoxide; echocardiography; intensive care
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: End tidal carbon monoxide — * Evaluation of cardiac output estimated by transthoracic echocardiography and end tidal carbon monoxide
  * Evaluation of cardiac output estimated by transthoracic echocardiography and portal veinous velocity
  * Evaluation of femoral veinous velocity
  Other Names: Transthoracic echocardiography

SUMMARY:
Hemodynamic monitoring, especially cardiac output assessment, is a key feature for the management of critically ill patients. Although the use of invasive methods, such as thermodilution with a pulmonary artery catheter, remains the GOLD standard for the evaluation of the cardiac output, several non-invasive techniques are currently used in practice. An acceptable estimation of the cardiac output can be made by standard transthoracic echocardiography. Cardiac output can be calculated from subaortic velocity time integral (VTI). However, this technique requires a trained operator and depends on the echogenicity of the patient. The best method for assessing cardiac output depends on the patient's needs, the clinical scenario and the physician's experience with the monitoring device itself. No simple and rapid tool currently exist for assessing cardiac output in critically ill patients.

The measurement of end-tidal carbon dioxide (EtCO2) used in routine in critically ill patients requiring mechanical ventilation could be an interesting alternative. Indeed, the amount of carbon dioxide (CO2) exhaled depends on the production of CO2 by the body, the pulmonary blood flow (corresponding to cardiac output) and its elimination by alveolar ventilation. In controlled ventilation, ie for constant alveolar ventilation, EtCO2 should therefore depend only on cardiac output. It has been shown in a porcine model that EtCO2 and cardiac output are strongly related under stable respiratory and metabolic conditions. In humans, only the variation of EtCO2 after volume expansion has been studied and EtCO2 seems to reflect changes in cardiac output. Nevertheless, the usefulness of EtCO2 in assessing cardiac output has never been evaluated.

The objective of this study is therefore to determine the relationship between EtCO2 and cardiac output evaluated by the measurement of subaortic VTI in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* patients intubated and ventilated in the control assisted mode with no inspiratory effort
* requiring vasopressors

Exclusion Criteria:

* less than 18 years
* refuse to participate
* situation in which health condition, medication or procedure could significantly interfere with the interpretation of EtCO2 or cardiac output (extracorporeal life support, pneumothorax with persistant air leak)

(be increased without correlation to an infectious process (poly-traumatised patients,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients > 18 years intubated and ventilated in the control assisted mode with no inspiratory effort referred to the intensive unit.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between cardiac output (VTI) and EtCO2 | between 0 to 3 day after ICU admission
  ITV ≈ (FR x EtCO2)/PaCO2

SECONDARY OUTCOMES:
Increase the sensitivity for detection of low cardiac output by using EtCO2 | between 0 to 3 day after ICU admission
  Estimate (development population) and validate (validation population) cut-off to detect low cardiac output by using EtCO2
Correlation between cardiac output (VTI) and portal veinous velocity | between 0 to 3 day after ICU admission
Comparison between cardiac output (VTI) and femoral veinous velocity | between 0 to 3 day after ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive care unit, University hospital of Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mercado P, Maizel J, Beyls C, Titeca-Beauport D, Joris M, Kontar L, Riviere A, Bonef O, Soupison T, Tribouilloy C, de Cagny B, Slama M. Transthoracic echocardiography: an accurate and precise method for estimating cardiac output in the critically ill patient. Crit Care. 2017 Jun 9;21(1):136. doi: 10.1186/s13054-017-1737-7. PMID 28595621
- [Background] Long B, Koyfman A, Vivirito MA. Capnography in the Emergency Department: A Review of Uses, Waveforms, and Limitations. J Emerg Med. 2017 Dec;53(6):829-842. doi: 10.1016/j.jemermed.2017.08.026. Epub 2017 Oct 7. PMID 28993038
- [Background] Weil MH, Bisera J, Trevino RP, Rackow EC. Cardiac output and end-tidal carbon dioxide. Crit Care Med. 1985 Nov;13(11):907-9. doi: 10.1097/00003246-198511000-00011. PMID 3931979
- [Background] Monnet X, Bataille A, Magalhaes E, Barrois J, Le Corre M, Gosset C, Guerin L, Richard C, Teboul JL. End-tidal carbon dioxide is better than arterial pressure for predicting volume responsiveness by the passive leg raising test. Intensive Care Med. 2013 Jan;39(1):93-100. doi: 10.1007/s00134-012-2693-y. Epub 2012 Sep 19. PMID 22990869